CLINICAL TRIAL: NCT05437848
Title: A Phase 1 Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Cotadutide in Chinese Overweight/Obese Subjects With Type 2 Diabetes Mellitus
Brief Title: Chinese Multiple Dose Escalation (MDE) High Dose Study
Acronym: COTA China PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5671C00005
Record Dates: First submitted 2022-02-23; First posted 2022-06-29 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Diabetes
Keywords: Diabetes; Cotadutide; MEDI0382; D5671C00005; Type 2 Diabetes mellitus; Obesity; Overweight
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Total 16 Chinese subjects will be randomized to cotadutide or placebo in a 3:1 ratio (cotadutide [n=12] and placebo [n=4]) at multicenter in China mainland.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cotadutide (Experimental): Those subjects who were randomized to cotadutide once daily SC will begin at 50 μg once daily, then up-titrated to 100 μg once daily a week later, after that up-titration will be done at 100 μg increment weekly, till to a maximum of 600 μg once daily.
  Interventions: Drug: Experimental: Cotadutide
- Placebo (Placebo Comparator): Placebo: Placebo subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Experimental: Cotadutide — Cotadutide: subcutaneous (SC) injection
  Arms: Cotadutide
Other: Placebo — Placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
A Phase 1 Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Cotadutide in Overweight/Obese Subjects with Chinese ancestry with Type 2 Diabetes Mellitus

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled study designed to evaluate the safety, tolerability, PK and efficacy of ascending doses of cotadutide in overweight or obese subjects with T2DM. This study will enroll subjects aged 18 to 74 years with a body mass index (BMI) ≥ 25 and ≤ 35 kg/m2. Subjects will have a diagnosis of T2DM and inadequate blood glucose control as defined by a HbA1c of 7% to 8.5%, and will be on metformin monotherapy in the three months prior to screening. Total 16 Chinese subjects will be randomized to cotadutide or placebo in a 3:1 ratio (cotadutide [n=12] and placebo [n=4]) at multicentre in China mainland. Those subjects who receive cotadutide once daily SC will be titrated to a maximum of 600 μg once daily SC, beginning at 50 μg once daily SC. The study has about 2 weeks screening period, a run-in period of 10 days and an up to 7-week up-titration treatment period followed by a 3-week treatment extension period at the dose of 600 μg and followed by a 28-day follow-up period.

ELIGIBILITY:
Inclusion Criteria

1. Subjects aged 18 to 74 years
2. Provision of signed and dated written informed consent prior to any study specific procedures
3. BMI between 25 and 35 kg/m2
4. HbA1c range of 7% to 8.5%
5. Willing and able to self-inject investigational product
6. Diagnosed with T2DM with glucose control managed with metformin monotherapy where no significant dose change has occurred in the three months prior to screening.
7. Women of child-bearing potential who are sexually active with a male partner must be using at least one highly effective method of contraception. And must have a negative serum or urine pregnancy test within 72 hours prior to the start of IP, and must not be breastfeeding.

Exclusion Criteria

1. Any subject who has received another IP as part of a clinical study or a GLP-1 analogue containing preparation within the last 30 days or 5 half-lives of the drug (whichever is longer) at the time of screening
2. Concurrent participation in another randomization study of any kind; repeat randomization is prohibited
3. Any subject who has received any of the following medications within the specified timeframe prior to the start of the study

   * Herbal preparations for control of body weight or appetite
   * Drugs licensed for control of body weight or appetite
   * Opiates, domperidone, metoclopramide, or other drugs known to alter gastric emptying
   * Antimicrobials within the quinolone (eg, ciprofloxacin), macrolide (eg, clarithromycin) or azole class (eg, ketoconazole)
   * Any change in antihypertensive medication
   * Aspirin (acetylsalicylic acid) at a dose greater than 150 mg once daily
   * Paracetamol (acetaminophen) or paracetamol-containing preparations at a total daily dose of greater than 3000 mg
   * Ascorbic acid (vitamin C) supplements at a total daily dose of greater than 1000 mg
4. Symptoms of acutely decompensated blood glucose control, recent severe hypoglycemia, a history of T1DM orDKA
5. Acute pancreatitis at screening or history of acute pancreatitis or chronic pancreatitis or serum triglyceride levels > 11 mmol/L at screening
6. Significant inflammatory bowel disease, gastroparesis or other severe disease or surgery affecting the upper GI tract, which may affect gastric emptying or could affect the interpretation of safety and tolerability data
7. Significant hepatic disease (except for NASH or NAFLD without portal hypertension or cirrhosis) and/or subjects with any of the following results at screening:

   * AST ≥ 3 × ULN
   * ALT ≥ 3 × ULN
   * TBL ≥ 2 × ULN
8. Impaired renal function defined as eGFR< 30 mL/minute/1.73m2 at screening
9. Poorly controlled hypertension defined as:

   * SBP > 160 mmHg
   * DBP or ≥ 90 mmHg - After 10 minutes of supine rest and confirmed by repeated measurement at screening. Subjects who fail BP screening criteria may be considered for 24-hour ABPM at the discretion of the investigator. Subjects who maintain a mean 24-hour BP < 160/100 mmHg with a preserved nocturnal dip of > 15% will be considered eligible.
10. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting 12-lead ECG or any abnormalities that may interfere with the interpretation of serial ECG changes, including QTc interval changes at screening, as judged by the investigator, and prolonged QTcF > 450 ms, or family history of long QT-segment at screening
11. PR (PQ) interval prolongation, intermittent second (Wenckebach block while asleep is not exclusive), or third-degree AV block, or AV dissociation
12. Persistent or intermittent complete bundle branch block.
13. Unstable angina pectoris, myocardial infarction, transient ischemic attack, or stroke within 3 months prior to screening, or subjects who have undergone percutaneous coronary intervention or a coronary artery bypass graft within the past 6 months or who are due to undergo these procedures at the time of screening
14. Severe congestive heart failure (NYHA Class III or IV)
15. Basal calcitonin level ≥ 50 ng/L at screening or history/family history of medullary thyroid carcinoma or MEN2
16. History of neoplastic disease within 5 years prior to screening, except for adequately treated basal cell, squamous cell skin cancer, or in situ cervical cancer
17. Any positive results for serum hepatitis B surface antigen, hepatitis C antibody, and HIV antibody
18. History of substance dependence, alcohol abuse, or excessive alcohol intake within 3 years prior to screening and/or a positive screen for drugs of abuse or alcohol at screening or on admission to the study unit.
19. Symptoms of depression or any other psychiatric disorder requiring treatment with medication (eg, anti-depressants, anti-psychotics) at screening. However, subjects who use benzodiazepines for chronic anxiety or sleep disorders may be permitted to enter the study.
20. History of severe allergy/hypersensitivity, including to any component of the investigational product formulation or other biological agent, or ongoing clinically important allergy/hypersensitivity as judged by the investigator
21. Blood/plasma donation within 1 month of screening
22. Involvement of any AstraZeneca, the contract research organization, or the virtual study site employee or their close relatives
23. For women only- currently pregnant (confirmed with positive pregnancy test) or breastfeeding

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Baseline until the follow-up period (28 days post last dose), 98 days in total
  To assess the safety and tolerability of Cotadutide
Incidence of treatment-emergent serious adverse events (TESAEs) | Baseline until the follow-up period (28 days post last dose), 98 days in total
  To assess the safety and tolerability of Cotadutide
Number of Participants With Abnormal Electrocardiograms (ECGs) Reported as TEAEs | Baseline until the follow-up period (28 days post last dose), 98 days in total
  Number of participants with abnormal ECGs reported as TEAEs are reported. Abnormal ECGs is defined as any abnormal findings in heart rate, RR interval, PR interval, QRS, QT intervals, and QTcF intervals as measured by digitial 12-lead ECG.
Number of participants with abnormal vital signs reported as TEAEs | Baseline until the follow-up period (28 days post last dose), 98 days in total
  Number of participants with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs are defined as any abnormal findings in the vital sign parameters (Systolic Blood Pressure, Diastolic Blood Pressure, Pulse, Respiration rate, body temperature).
Number of Participants With Abnormal Physical Examinations Reported as TEAEs | Baseline until the follow-up period (28 days post last dose), 98 days in total
  Number of participants with abnormal physical examinations reported as TEAEs are reported. Abnormal physical examinations findings are defined as any abnormal finding in the following body systems: immunologic/allergy; head, ears, eyes, nose and throat; respiratory; cardiovascular; gastrointestinal; musculoskeletal; neurological psychiatric; dermatologic; hematologic/lymphatic; and enocrine.
Area under the concentration-time curve (AUC) during the dosing interval (AUCtau) | Day 1 of Up-titration treatment period through 3 days post lost dose, total of up to 73 days.
  To characterize the PK profile of Cotadutide
Maximum observed concentration (Cmax) | Day 1 of Up-titration treatment period through 3 days post lost dose, total of up to 73 days.
  To characterize the PK profile of Cotadutide
Time to Cmax (tmax) | Day 1 of Up-titration treatment period through 3 days post lost dose, total of up to 73 days.
  To characterize the PK profile of Cotadutide
Trough plasma concentration (Ctrough) | Day 1 of Up-titration treatment period through 3 days post lost dose, total of up to 73 days.
  To characterize the PK profile of Cotadutide
Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs | Baseline until the follow-up period (28 days post last dose), 98 days in total
  Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs are reported. Abnormal clinical laboratory parameters defined as any abnormal finding during analysis of serum chemistry, hematology, and urinalysis.

SECONDARY OUTCOMES:
Anti-drug antibodies (ADAs) to Cotadutide | Day 1 of Up-titration treatment period through end of study, 98 days in total
  To characterize the immunogenicity of Cotadutide
Change in daily average glucose levels | baseline to the end of extension period, and during 14 days of the follow up period, 84 days in total.
  To assess the effect of Cotadutide on glucose control as measured by continuous glucose monitoring (CGM)
Change in 7-day average glucose levels | Baseline (Days -7 to -1), Days 1-7, Days 8-14, Days 15-21, Days 22-28, Days 29-35, Days 36-42, Days 43-49 of the up-titration period, Days 50-56, Days 57-63, Days 64 - 70 of the treatment extension period
  To assess the effect of Cotadutide on glucose control as measured by continuous glucose monitoring (CGM)
Change in percentage time spent in hyperglycemia (> 140 mg/dL) over 24hours and over 7days | Baseline (Days -7 to -1), Days 1-7, Days 8-14, Days 15-21, Days 22-28, Days 29-35, Days 36-42, Days 43-49 of the up-titration period, Days 50-56, Days 57-63, Days 64 - 70 of the treatment extension period
  To assess the effect of Cotadutide on glucose control as measured by continuous glucose monitoring (CGM)
Change in percentage time spent in target range (70 -140 mg/dL) over 24hours and over 7days | Baseline (Days -7 to -1), Days 1-7, Days 8-14, Days 15-21, Days 22-28, Days 29-35, Days 36-42, Days 43-49 of the up-titration period, Days 50-56, Days 57-63, Days 64 - 70 of the treatment extension period
  To assess the effect of Cotadutide on glucose control as measured by continuous glucose monitoring (CGM)
Change in percentage time spent in the range (< 54 mg/dL) over 24hours and over 7days | Baseline (Days -7 to -1), Days 1-7, Days 8-14, Days 15-21, Days 22-28, Days 29-35, Days 36-42, Days 43-49 of the up-titration period, Days 50-56, Days 57-63, Days 64 - 70 of the treatment extension period
  To assess the effect of Cotadutide on glucose control as measured by continuous glucose monitoring (CGM)
Change in estimated hemoglobin A1c (HbA1c) | Baseline through 21day treatment extension period, 70 days in total
  To assess the effect of Cotadutide on glucose control as measured by continuous glucose monitoring (CGM)
Change in fasting plasma glucose (mg/dL) | Baseline through 21day treatment extension period, 70 days in total
  To assess the effects of cotadutide, titrated up to the dose of 600 μg, on additional measures of glucose control
Change in HbA1c | Baseline through 21day treatment extension period, 70 days in total
  To assess the effects of cotadutide, titrated up to the dose of 600 μg, on additional measures of glucose control
Percentage change in body weight | Baseline through 21day treatment extension period, 70 days in total
  To assess the effects of cotadutide, titrated up to the dose of 600 μg, on body weight
Absolute change in body weight | Baseline through 21day treatment extension period, 70 days in total
  To assess the effects of cotadutide, titrated up to the dose of 600 μg, on body weight
Proportion of subjects achieving > 5% body weight loss | Baseline through 21day treatment extension period, 70 days in total
  To assess the effects of cotadutide, titrated up to the dose of 600 μg, on body weight
Change in coefficient of variation as measured by CGM over 7 days | Baseline (Days -7 to -1), Days 1-7, Days 8-14, Days 15-21, Days 22-28, Days 29-35, Days 36-42, Days 43-49 of the up-titration period, Days 50-56, Days 57-63, Days 64 - 70 of the treatment extension period
  To assess the effect of Cotadutide on glucose control as measured by continuous glucose monitoring (CGM)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Research Site, Guangzhou
  - Research Site, Nanjing

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home